CLINICAL TRIAL: NCT01277692
Title: A Randomized, Double Blind, Dose Escalation, Fusion, First Time in Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Single and Repeat Doses of GSK2336805 in Healthy Volunteers and Single Doses in Chronically Infected Hepatitis C Subjects
Brief Title: A First Time in Human Study to Assess GSK2336805 in Healthy Volunteers and Single Doses in Chronically Infected Hepatitis C Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 114885
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis C
Keywords: First administration to human, safety, pharmacokinetics, healthy subjects, antiviral activity, hepatitis C patients
MeSH Terms: conditions — Hepatitis C | interventions — GSK2336805

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: Single Dose Escalation in Healthy Subjects (Experimental): The doses currently planned are 10, 30mg, 100mg, 200mg
  Interventions: Drug: GSK2336805 10mg; Drug: GSK2336805 30mg; Drug: GSK2236805 100mg; Drug: GSK2236805 200mg
- Part 2: Repeat Dose Escalation in Healthy Subjects (Experimental): The first planned dose is currently 10mg QD and the planned maximum dose is 100mg QD
  Interventions: Drug: GSK2236805 10mg; Drug: GSK2236805 dose to be determined up to 100mg
- Part 3: Single Dose Escalation in HCV Infected Subjects (Experimental): The planned doses for Part 3 are 5mg, 30mg, and 100 mg.
  Interventions: Drug: GSK2236805 5mg; Drug: GSK2236805 30mg; Drug: GSK2236805 100mg

INTERVENTIONS:
Drug: GSK2336805 10mg — single dose once daily
  Arms: Part 1: Single Dose Escalation in Healthy Subjects
Drug: GSK2336805 30mg — single dose once daily
  Arms: Part 1: Single Dose Escalation in Healthy Subjects
Drug: GSK2236805 100mg — single dose once daily
  Arms: Part 1: Single Dose Escalation in Healthy Subjects
Drug: GSK2236805 200mg — single dose once daily
  Arms: Part 1: Single Dose Escalation in Healthy Subjects
Drug: GSK2236805 10mg — repeat dose once daily for 7 days
  Arms: Part 2: Repeat Dose Escalation in Healthy Subjects
Drug: GSK2236805 dose to be determined up to 100mg — repeat dose once daily for 7 days
  Arms: Part 2: Repeat Dose Escalation in Healthy Subjects
Drug: GSK2236805 5mg — single dose in HCV infected patients
  Arms: Part 3: Single Dose Escalation in HCV Infected Subjects
Drug: GSK2236805 30mg — single dose in HCV infected patients
  Arms: Part 3: Single Dose Escalation in HCV Infected Subjects
Drug: GSK2236805 100mg — single dose in HCV infected patients
  Arms: Part 3: Single Dose Escalation in HCV Infected Subjects

SUMMARY:
This study is a three Part, Phase 1, randomized, dose-escalation, fusion, placebo-controlled, double-blind study to determine the safety, tolerability and Pharmacokinetic (PK) profile of GSK2336805 in healthy subjects and the safety, tolerability, PK, and antiviral profile of GSK2336805 in subjects chronically infected with HCV: i. Single doses in healthy subjects and the effect of food on GSK2336805 PK (Part 1). ii. Repeat doses in healthy subjects (Part 2) iii. Single doses in chronically infected HCV positive subjects (Part 3).

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG, including no cardiac, pulmonary, hepatic, biliary (except Gilbert's disease, gastrointestinal, or renal (defined as serum creatinine >1.5 mg/dL or a calculated creatinine clearance (CrCl)<50 mL/min), disorders, or cancer within the past 5 years (except localized or in situ cancer of the skin). A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. A single repeat laboratory evaluation is allowed for eligibility determination.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female is eligible to enter and participate in this study if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, bilateral oophorectomy, hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea.
* Male subjects must agree to use one of the contraception methods listed in the protocol.
* Body weight greater than or equal to 50 kg (110 lbs.) for men and greater than or equal to 45 kg (99 lbs.) for women. For Part 1, body mass index (BMI) between 18.5-32 kg/m2 inclusive will be allowed. For Part 3, BMI between 18.5-35.0 kg/m2 inclusive will be allowed.
* For healthy subjects in Part 1 and Part 2, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase, bilirubin, and creatinine less than the upper limits of normal (ULN) (isolated bilirubin <2.0xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QTcB or QTcF < 450 msec; or QTc <480 msec in subjects with Bundle Branch Block.
* The subject's systolic blood pressure is inside the range of 90-140 mmHg, or diastolic blood pressure is inside the range of 45-90 mmHg or heart rate is inside the range of 50-100 beats per minute (bpm) for female subjects or 45-100 bpm for male subjects.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned.
* The following are Supplemental inclusion criteria for Part 3: HCV positive subjects: Treatment naive chronically infected genotype 1 HCV patients, defined as infection for >6 months and no prior HCV therapy.
* An HCV RNA viral load of greater than 100,000 IU/mL using a COBAS TaqMan HCV test and HCV genotype 1a or 1b as assessed by VERSANT HCV genotyping LiPA 2.0 (Bayer Healthcare, Berkeley, California), or by direct Deoxyribonucleic acid (DNA) sequencing of the NS5B gene Hepatitis C virus infection of mixed genotype excluded. HCV subjects with mixed genotypes are not eligible for the study.
* ALT greater than or equal to 3x ULN is allowed.
* Liver biopsy within two years prior to screening indicating the absence of cirrhosis.

Exclusion Criteria:

* Unwillingness or inability to follow the procedures outlined in the protocol.
* A positive pre-study test for Human Immunodeficiency Virus (HIV) antibody or Hepatitis B surface antigen.
* For healthy subjects in Parts 1 and 2, a positive Hepatitis C antibody result within 3 months of screening. Chronic HCV infected subjects in Part 3 will have a positive HCV antibody and a positive HCV RNA.
* Pregnant females as determined by positive serum or urine Human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Subject is mentally or legally incapacitated.
* Has a history of regular alcohol consumption averaging: >7 drinks/week for women or >14 drinks/week for men within 6 months of the screening visit.
* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* For healthy subjects in Parts 1 and 2, history of regular use of tobacco- or nicotine-containing products within 3 months of the screening visit or indication of tobacco use as evidenced by a positive urine cotinine test at screening. For chronic HCV infected subjects in Part 3, history of regular use of tobacco- or nicotine-containing products is allowed; however, use of tobacco is not allowed on days of PK draws nor at the study site.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, satsuma, ugli, tangerine, and tangelo, exotic citrus fruits, grapefruit hybrids or fruit juices from 5 days prior to the first dose of study medication.
* The subject has a positive pre-study drug screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids, phencyclidine (PCP), and benzodiazepines. Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new investigational entities within 12 months prior to the first dosing day.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Holter monitoring shows one or more of the following: Any symptomatic arrhythmia (except isolated extra systoles); Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, sustained ventricular tachycardia (SVT) (>10 consecutive beats)); Non-sustained or sustained ventricular tachycardia (defined as >3 consecutive ventricular ectopic beats); Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree or higher in an awake subject], Wolff-Parkinson-White syndrome (WPW) syndrome, other pre-excitation syndromes); Symptomatic sinus pause or sinus pause >3 seconds - unless patient is straining, vomiting, or having some other type of hypervagal response; 300 or more supraventricular ectopic beats in 24 hours; 250 or more ventricular ectopic beats in 24 hours; Ischemia, diagnosed by a sequence of EKG changes that include flat or down sloping ST-segment depression >0.1 mV, with a gradual onset and offset that lasts for a minimum period of 1 minute. Each episode of ischemia must be separated by a minimum duration of at least 1 minute, during which the ST segment returns back to baseline (1x1x1 rule)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-11-03 (Actual); Primary Completion 2011-05-09 (Actual); Study Completion 2011-05-09 (Actual)

PRIMARY OUTCOMES:
GSK2336805 safety parameters : adverse events | Part 1 change from baseline for 14 days; Part 2 change from baseline for 24 days; Part 3 change from baseline for 16 days
GSK2336805 safety parameters: telemetry | Part 1 change from baseline for 14 days; Part 2 change from baseline for 24 days; Part 3 change from baseline for 16 days
GSK2336805 safety parameters: absolute values and changes over time of hematology, clinical chemistry, urinalysis | Part 1 change from baseline for 14 days; Part 2 change from baseline for 24 days; Part 3 change from baseline for 16 days
GSK2336805 safety parameters: vital signs (blood pressure, heart rate) | Part 1 change from baseline for 14 days; Part 2 change from baseline for 24 days; Part 3 change from baseline for 16 days
GSK2336805 safety parameters: electrocardiogram (ECG) parameters | Part 1 change from baseline for 14 days; Part 2 change from baseline for 24 days; Part 3 change from baseline for 16 days
GSK2336805 PK parameters following single dose administration: area under the plasma concentration curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity) | Part 1 up to 48 hours; Part 2 for 7 and 14 days; Part 3 for 48 hours
GSK2336805 PK parameters following single dose administration: area under the plasma concentration curve over the dosing interval AUC(0-tau)) | Part 1 up to 48 hours; Part 2 for 7 and 14 days; Part 3 for 48 hours
GSK2336805 PK parameters following single dose administration: maximum observed concentration (Cmax) | Part 1 up to 48 hours; Part 2 for 7 and 14 days; Part 3 for 48 hours
GSK2336805 PK parameters following single dose administration: time to maximum observed concentration (tmax) | Part 1 up to 48 hours; Part 2 for 7 and 14 days; Part 3 for 48 hours
GSK2336805 PK parameters following single dose administration: observed concentration at 24h post-dose (C24) | Part 1 up to 48 hours; Part 2 for 7 and 14 days; Part 3 for 48 hours
GSK2336805 PK parameters following single dose administration: terminal half-life (t1/2) | Part 1 up to 48 hours; Part 2 for 7 and 14 days; Part 3 for 48 hours
GSK2336805 PK parameters following single dose administration: lag time (tlag) | Part 1 up to 48 hours; Part 2 for 7 and 14 days; Part 3 for 48 hours
GSK2336805 PK parameters following single dose administration: apparent clearance (CL/F) | Part 1 up to 48 hours; Part 2 for 7 and 14 days; Part 3 for 48 hours
GSK2336805 PK parameters following repeat dose administration:AUC(0-tau) | Day 7 and Day 14
GSK2336805 PK parameters following repeat dose administration: Pre-dose (trough) concentration at the end of the dosing interval Ctau | Day 7 and Day 14
GSK2336805 PK parameters following repeat dose administration: Cmax | Day 7 and Day 14
GSK2336805 PK parameters following repeat dose administration: tmax | Day 7 and Day 14
GSK2336805 PK parameters following repeat dose administration: t1/2, | Day 7 and day 14
GSK2336805 PK parameters following repeat dose administration: CL/F | Day 7 and Day 14
GSK2336805 PK parameters following single dose in HCV infected subjects: AUC(0-infinity) or AUC(0 - tau) | for 48 hours
GSK2336805 PK parameters following single dose in HCV infected subjects: Cmax | for 48 hours
GSK2336805 PK parameters following single dose in HCV infected subjects: C24 | for 48 hours
GSK2336805 PK parameters following single dose in HCV infected subjects: tmax | for 48 hours
GSK2336805 PK parameters following single dose in HCV infected subjects: tlag | for 48 hours
GSK2336805 PK parameters following single dose in HCV infected subjects: CL/F | for 48 hours
HCV Ribonucleic acid (RNA) viral load reduction from baseline during the 24hr and post-dosing following a single dose of GSK2336805 in HCV subjects | at baseline, 24 hours, and for 16 days
HCV RNA change from baseline to nadir (maximum change) in HCV subjects | baseline, and for 16 days
Time course of HCV viral load at baseline, after dosing with GSK2336805, and for greater than or equal to 2 weeks after GSK2336805 dosing (Part 3) | baseline and up to 16 days

SECONDARY OUTCOMES:
GSK2336805 PK parameters: AUC(0-infinity) or AUC (0 - tau) following single dose administration of a given dose of GSK2336805 with and without moderate fat/calorie meal (Part 1) | 48 hours
GSK2336805 PK parameters: Cmax following single dose administration of a given dose of GSK2336805 with and without moderate fat/calorie meal (Part 1) | 48 hours
GSK2336805 PK parameters: tmax following single dose administration of a given dose of GSK2336805 with and without moderate fat/calorie meal (Part 1) | 48 hours
GSK2336805 PK parameters: tlag following single dose administration of a given dose of GSK2336805 with and without moderate fat/calorie meal (Part 1) | 48 hours
GSK2336805 AUC(0-tau) on Day 7 compared to AUC(0-24) on Day 1 to estimate accumulation ratio (R) and GSK2336805 AUC(0-tau) on Day 7 compared to AUC(0-infinity) on Day 1 | Day 1 and Day 7
Pre-dose concentrations (Ctau) on Day 2 through 7 to assess the achievement of steady state of GSK2336805 following repeat administration (Part 2) | Day 2 through Day 7
GSK2336805 PK parameters: AUC(0-infinity), AUC(0-t), Cmax, and C24 following single dose administration | 48 hours
GSK2336805 PK parameters: AUC(0-τ), Cτ, and Cmax following repeat administration | for 7 days
Correlation between concentration and various safety parameters, if appropriate | 16 days
Sequence analysis of the viral quasispecies as appropriate (Part 3). | 16 days
GSK2336805 AUC(0-tau) on Day 14 compared to AUC(0-24) on Day 1 to estimate accumulation ratio (R) and GSK2336805 AUC(0-tau) on Day 14 compared to AUC(0-inf) on Day 1 | 14 days
Pre-dose concentrations (Ctau) on Day 2 through 14 to assess the achievement of steady state of GSK2336805 following repeat administration (Part 2 Cohort E) | Day 2 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Willingboro, New Jersey

REFERENCES:
- [Background] Wilfret DA, Walker J, Adkison KK, Jones LA, Lou Y, Gan J, Castellino S, Moseley CL, Horton J, de Serres M, Culp A, Goljer I, Spreen W. Safety, tolerability, pharmacokinetics, and antiviral activity of GSK2336805, an inhibitor of hepatitis C virus (HCV) NS5A, in healthy subjects and subjects chronically infected with HCV genotype 1. Antimicrob Agents Chemother. 2013 Oct;57(10):5037-44. doi: 10.1128/AAC.00910-13. Epub 2013 Jul 29. PMID 23896477
- See also: Results for study 114885 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114885?search=study&search_terms=114885#rs